CLINICAL TRIAL: NCT06445361
Title: The Prevalence of Non-Alcoholic Fatty Liver Disease in Type 1 Diabetes Mellitus Patients Followed at Ziekenhuis Oost-Limburg, Genk, Belgium
Brief Title: Prevalence of NAFLD in T1DM Patients
Acronym: PAD1ZOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Z-2022007
Record Dates: First submitted 2024-02-28; First posted 2024-06-06 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: NAFLD; Type 1 Diabetes; Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study cohort (Other): FibroScan measurement
  Interventions: Diagnostic Test: FibroScan

INTERVENTIONS:
Diagnostic Test: FibroScan — Performance of a FibroScan measurement to determine steatosis and fibrosis.

SUMMARY:
To determine the prevalence of NAFLD in T1DM patients.

ELIGIBILITY:
Inclusion Criteria:

* T1DM
* ≥ 18 years of age
* Written informed consent obtained

Exclusion Criteria:

* Excessive alcohol use
* Exclusion of other causes of liver disease and secondary causes of liver steatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NAFLD in T1DM | During the intervention
  To determine the prevalence of steatosis in a cohort of T1DM patients followed at the Departments of Endocrinology in ZOL by means of the FibroScan® device with controlled attenuation parameter (CAP) measurements.
Prevalence of fibrosis in T1DM | During the intervention
  To determine the prevalence of fibrosis in a cohort of T1DM patients followed at the Departments of Endocrinology in ZOL by means of the FibroScan® device with vibration controlled attenuation parameter (VCTE) measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No
During the study period IPD will not be made available for other researchers. When the study is completed and results are reported, IPD can be shared.